CLINICAL TRIAL: NCT05355649
Title: Impact of a New Aspiration Technique-based Device for Assessment of Cervical Stiffness in Pregnant Women With Symptoms of Preterm Labour
Brief Title: Aspiration Technique-based Device for Preterm Labor
Acronym: PREGNOLIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal investigator, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VanvFedII
Record Dates: First submitted 2022-04-10; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Preterm Labor; Preterm Birth
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Intervention Model Description: PREGNOLIA SYSTEM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PREGNOLIA TEST (Other): Women at the time of triage will be tested with TVU CL (transvaginal ultrasound cervical length) and with the PREGNOLIA system
  Interventions: Device: PREGNOLIA SYSTEM

INTERVENTIONS:
Device: PREGNOLIA SYSTEM — The Pregnolia System is composed of two products: an active device (Pregnolia Control Unit) and a single-use sterile probe (Pregnolia Probe).
  The intended use of the Pregnolia System is to provide information about the mechanical properties of the uterine cervix by assessing the tissue stiffness through a proxy parameter (the closing pressure, denominated CSI, or Cervical Stiffness Index, in mbar). The Pregnolia System is intended to be used in conjunction with the information obtained from the clinical evaluation of the patient and in addition to other standard examinations.

SUMMARY:
Premature birth (PTB, birth before 37 weeks of pregnancy) is a global, yet unsolved, problem. With a global amount of approximately 15 M babies born prematurely, PTB is the leading cause of perinatal morbidity and mortality in many countries. Furthermore, premature babies often have complicated medical problems, especially those born very early.

Some women spontaneously deliver prematurely without any symptom or sign of the imminent labor, whereas others present with symptoms of preterm labor (PTL). In the latter case, clinicians can intervene and treat the woman with tocolytics and antenatal corticosteroids in order to accelerate fetal lung maturation and reduce the risk of respiratory distress syndrome. However, one of the major challenges in the management of women presenting with symptoms of PTL is to distinguish between true and false PTL with the existing clinical methods (digital examination or transvaginal cervical length assessment). In fact, over 50% of the women presenting with PTL symptoms do not deliver prematurely and are still unnecessarily hospitalized and treated with corticosteroids as well as tocolytics, and only less than 10% of women give birth within 7 days of presentation. Unnecessary treatments and hospitalizations also result in increased health costs.

Thus, there is a need for more accurate methods and tools to evaluate the cervical maturation status as indication of imminent labor in order to avoid unnecessary hospital admissions and therapy.

Recently, cervical stiffness has been evaluated as more reliable tool for prediction of spontaneous preterm birth. Cervical stiffness can be evaluated using ultrasound by cervical elastography , but also by an aspiration technique-based method with a novel CE-marked device, the Pregnolia System.

Thus, the aims of this study are to evaluate:

* if the cervical stiffness measured with the Pregnolia System can differentiate between women with true PTL and those with false PTL,
* if the knowledge of cervical stiffness improves the detection of women at true risk of spontaneous preterm birth in combination or over state of the art (e.g. cervical length on TVUS).

DETAILED DESCRIPTION:
Premature birth (PTB, birth before 37 weeks of pregnancy) is a global, yet unsolved, problem. With a global amount of approximately 15 M babies born prematurely, PTB is the leading cause of perinatal morbidity and mortality in many countries. Furthermore, premature babies often have complicated medical problems, especially those born very early.

Some women spontaneously deliver prematurely without any symptom or sign of the imminent labor, whereas others present with symptoms of preterm labor (PTL). In the latter case, clinicians can intervene and treat the woman with tocolytics and antenatal corticosteroids in order to accelerate fetal lung maturation and reduce the risk of respiratory distress syndrome. However, one of the major challenges in the management of women presenting with symptoms of PTL is to distinguish between true and false PTL with the existing clinical methods (digital examination or transvaginal cervical length assessment). In fact, over 50% of the women presenting with PTL symptoms do not deliver prematurely and are still unnecessarily hospitalized and treated with corticosteroids as well as tocolytics, and only less than 10% of women give birth within 7 days of presentation. Unnecessary treatments and hospitalizations also result in increased health costs.

Thus, there is a need for more accurate methods and tools to evaluate the cervical maturation status as indication of imminent labor in order to avoid unnecessary hospital admissions and therapy.

Recently, cervical stiffness has been evaluated as more reliable tool for prediction of spontaneous preterm birth. Cervical stiffness can be evaluated using ultrasound by cervical elastography , but also by an aspiration technique-based method with a novel CE-marked device, the Pregnolia System.

Thus, the aims of this study are to evaluate:

* if the cervical stiffness measured with the Pregnolia System can differentiate between women with true PTL and those with false PTL,
* if the knowledge of cervical stiffness improves the detection of women at true risk of spontaneous preterm birth in combination or over state of the art (e.g. cervical length on TVUS).

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestations with symptoms of preterm labor
* Gestational age between 24 and 33 weeks
* Maternal age ≥18 years

Exclusion Criteria:

* Cervical dilatation ≥ 3 cm;
* Rupture of membranes;
* Cerclage or pessary in place;
* Severe vaginal bleeding;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Value of the system in women with symptoms of preterm labor | up to 34 weeks
  detection rate of PREGNOLIA system in women with symptoms of preterm labor (sensitivity, specificity, detection rate).

SECONDARY OUTCOMES:
Birth outcomes | up to 34 weeks
  Correlation between the system of the results and birth outcome (gestational age at birth, time to delivery, mode of delivery)
Comparison between pregnolia system and cevical length | up to 34 weeks
  Detection rate of the two systems
the change of the calcaneus stiffness index (CSI) at triage and discharge | up to 34 weeks
  to determine the change of the CSI at triage and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Saccone, md, Principal Investigator — federico ii
Locations (1):
- Gabriele Saccone, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not planned yet

REFERENCES:
- [Derived] Colacurci D, Saccone G, Ammendola A, Buonomo G, Murolo C, Locci M. Cervical Stiffness Index as predictor of preterm birth in women with threatened preterm labor. Eur J Obstet Gynecol Reprod Biol. 2025 Dec 23;318:114910. doi: 10.1016/j.ejogrb.2025.114910. Online ahead of print. PMID 41456565